CLINICAL TRIAL: NCT00833209
Title: Orbitofrontal Cortex (OFC) Influence on Addictive Behaviour in Medication Overuse Headache (MOH) Deriving From Migraine
Brief Title: Orbitofrontal Cortex (OFC) Influence on Addictive Medication Overuse Headache (MOH) Deriving From Migraine
Acronym: MOH-PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2008/28
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Medication Overuse Headache
Keywords: Orbitofrontal cortex; Medication Overuse Headache; Chronic headache; withdrawal
MeSH Terms: conditions — Headache Disorders, Secondary; Headache Disorders | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Patients with Medication Overuse Headache (MOH)
  Interventions: Procedure: PET (withdrawal)
- 2 (Sham Comparator): controls suffering from migraine
  Interventions: Procedure: Imaging
- 3 (Sham Comparator): controls without any neurological disease
  Interventions: Procedure: Imaging

INTERVENTIONS:
Procedure: PET (withdrawal) — 3 (18F)FDG-PET (before withdrawal, 3 months, 1 year), 2 MRI (before withdrawal, 1 year), will take the Iowa Gambling Task Test(before withdrawal) and will answer questionnaires measuring psychological dimensions (before withdrawal, 3 months, 1 year)
  Arms: 1
Procedure: Imaging — 2 MRI (inclusion, 1 year) ; Iowa Gambling Task Test(inclusion) and questionnaires (inclusion)
  Arms: 2
Procedure: Imaging — 1 MRI ; Iowa Gambling Task test and questionnaires.
  Arms: 3

SUMMARY:
Medication Overuse Headache (MOH) is an illness affecting about 1,5 % of the general population. It is characterized by chronic headache occurring for at least 15 days a month, by a use of antimigraine drugs during at least 3 months for more than 10 days a month (for ergots, triptans, opiate derivates and combined analgesics) or for more than 15 days a month (for simple analgesics). The chronic headache must have occurred during the period of antimigraine drug abuse and the headache must have returned to its episodical pattern after withdrawal of antimigraine drugs. But, about 50% of the MOH patients will relapse during the first year following the antimigraine drugs withdrawal.

The pathophysiology of MOH is still largely unknown, and the role of antimigraine drug abuse in the transformation from migraine through MOH is not fully understood.

DETAILED DESCRIPTION:
We recently explored cerebral metabolism in these MOH patients using (18F)FDG-PET (Fluoro Dexoxy Glucose Positon Emission Tomography) comparing them with controls. Results showed a hypometabolism in the OFC, which persist immediately after the antimigraine drugs withdrawal. A similar pattern is observed in varied substance related disorders and should be a marker of addictive behaviour. It can be linked with difficulties in the decision-making process, which can be explored by the Iowa Gambling Task (IGT) test.

Several questions are still unanswered. What will this abnormality become in the long term ? Is it predictive of susceptibility for relapse? Can it be linked to a specific psychological profile (addictive behaviour)?

ELIGIBILITY:
Inclusion Criteria for patients :

* older than eighteen years
* suffering from MOH (ICHD-II criteria)
* French speaking
* who wish to go on a withdrawal procedure

Exclusion Criteria :

* pregnant women or women of child bearing age who are not using contraception
* post traumatic headaches
* illnesses interfering with the central nervous system functionning
* psychotic disorder or current major depressive episode
* contraindication for PET or MRI (Magnetic Resonnance Imaging)
* contraindication for all prophylactic treatment for migraine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
basal cerebral metabolism using (18F)FDG-PET | before withdrawal, 3 months, 1 year

SECONDARY OUTCOMES:
Relapse | All study long
Magnetic Resonance Imaging data | before withdrawal and at one year

CONTACTS AND LOCATIONS:
Overall Officials: Françoise RADAT, MD, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - C.H.U. de Bordeaux - Groupe Hospitalier Pellegrin - Service Médecine nucléaire, Bordeaux
  - CHU de Bordeaux - Hôpital Tastet Girard Centre Anti douleur, Bordeaux

REFERENCES:
- [Derived] Meyer M, Di Scala G, Edde M, Dilharreguy B, Radat F, Allard M, Chanraud S. Brain structural investigation and hippocampal tractography in medication overuse headache: a native space analysis. Behav Brain Funct. 2017 Apr 8;13(1):6. doi: 10.1186/s12993-017-0124-5. PMID 28390437